CLINICAL TRIAL: NCT02132130
Title: A Three-part, Multicenter, Open Label, Single Dose Study to Assess the Safety, Tolerability, and Efficacy of Intra Labyrinthine (IL) CGF166 in Patients With Severe-to-profound Hearing Loss
Brief Title: Safety, Tolerability and Efficacy for CGF166 in Patients With Unilateral or Bilateral Severe-to-profound Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCGF166X2201
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2021-03-30 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Unilateral Severe to Profound Hearing Loss OR Bilateral Severe to Profound Hearing Loss
Keywords: gene therapy; unilateral hearing loss; bilateral hearing loss; balance; vestibular; cochlear implant; hearing restoration
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CGF166 dose 20 uL (Experimental): single dose volume #1
  Interventions: Drug: CGF166
- CGF166 dose 30 and 40 uL (Experimental): single dose volume #2
  Interventions: Drug: CGF166
- CGF166 dose 40 uL (Experimental): single dose volume #3
  Interventions: Drug: CGF166
- CGF166 dose 60 uL (Experimental): single dose volume #4
  Interventions: Drug: CGF166
- CFG166 dose 30 uL (Experimental): Single dose volume #5
  Interventions: Drug: CGF166

INTERVENTIONS:
Drug: CGF166 — CGF166 is a recombinant adenovirus 5 (Ad5) vector containing the human Atonal transcription factor (Hath1) cDNA for administration via intra-labyrinthine infusion

SUMMARY:
The goal of the study was to evaluate the safety, tolerability, and the potential ability of CGF166 delivered through IL-infusion to improve hearing. CGF166 is a recombinant adenovirus 5 (Ad5) vector containing a cDNA encoding the human Atonal transcription factor (Hath1).

DETAILED DESCRIPTION:
This study evaluated the safety, tolerability, and potential efficacy of CGF166 and the associated delivery procedures in patients with severe-to-profound unilateral or bilateral hearing loss. Eligible patients were required to have documented, non-fluctuating hearing loss.

ELIGIBILITY:
For all Parts A, B and C of the study,

Inclusion criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. For all Parts A, B and C of the study, male or female patients, 18 to 75 years old, inclusive, with severe-to-profound bilateral hearing loss or unilateral hearing loss with intact vestibular function in the nonoperative ear. Non-fluctuating severe-to-profound hearing loss is required for the study ear and is defined as:

   * PTA within 10 dB of the PTA obtained at least 11 months previously.
   * Word recognition within 20% of previous test at least 11 months previously
3. Candidate ear ("study ear"): Minimal residual hearing based on the pure tone average of 0.5, 1, 2, and 4 kHz thresholds of ≤110 dB HL
4. Candidate ear ("study ear"): Pure tone audiometric thresholds of ≥50 dB HL for each testable octave frequency of 0.125 and 0.250 kHz, ≥70 dB HL for each testable octave frequency from 0.5 through 8 kHz and sentence recognition scores ≤50% at screening.

6. Patients with intact vestibular function in at least one ear (non-study ear) as measured by vestibular evoked myogenic potential (VEMP) 7. Able to communicate well with the investigator, to understand and comply with the requirements of the study 8. MRI scan within 6 months or at screening to confirm suitability for inner ear surgery 9. Patients must weigh at least 40 kg to participate in the study, and must have a body mass index (BMI) <45 kg/m2. BMI = Body weight (kg) / [Height (m)]2

Exclusion Criteria:

1. Patients with hearing loss caused by genetic/developmental disorders, e.g., cochlea aplasia
2. Patients with existing conductive hearing loss or mixed hearing loss as judged by the Principal Investigator following a thorough review of all of the trial hearing assessments;
3. Patients with a history of cochlear implant in the study ear
4. Hearing loss due to any other cause that would not be expected to respond to hair cell regeneration, for example mechanical trauma or central auditory lesions or lack of an auditory nerve
5. Patients who will require ototoxic drugs as routine therapy over the course of the study, for example cystic fibrosis patients
6. Any contraindication to the planned surgery or anesthesia as determined by the surgeon or anesthesiologist
7. Previous surgery in the study ear
8. Any otological history, such as chronic otitis, cholesteatoma, tympanic membrane perforation, that suggests poor candidacy for cochlear implant or inner ear surgery or suggests potential interference with study auditory or vestibular function tests
9. Pregnant women
10. Abnormal vital signs and/or ECG that suggest potential contraindication for planned study anesthesia
11. Past serious adverse reaction to anesthesia
12. Meniere's Disease
13. History of radiation therapy to the head and neck
14. Participation in a clinical trial within the last 30 days
15. Immunocompromised patients, as judged by the investigators based on patient history, physical exam and CBC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Plontke SK. Otology Jubilee: 150 years of the Archiv fur Ohrenheilkunde "Where do we come from?--Where are we?--Where are we going?". Eur Arch Otorhinolaryngol. 2015 Jun;272(6):1301-3. doi: 10.1007/s00405-015-3538-4. Epub 2015 Feb 18. No abstract available. PMID 25690605
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 subjects were enrolled in the study, of which 19 completed the study and 2 subjects discontinued due to lost to follow-up and 1 subject withdrew consent
Pre-assignment Details: Safety analysis set comprised all subjects who received study drug and with no protocol deviations having relevant impact on safety.
Groups:
- CGF166 Dose 20 μL: single dose volume #1
- CGF166 Dose 30 μL: single dose volume #2
- CGF166 Dose 40 μL: single dose volume #3
- CGF166 Dose 60 μL: single dose volume #4
Period: Overall Study
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL
Started | 3 | 12 | 4 | 3
Completed | 3 | 10 | 4 | 2
Not Completed | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 3 | 2 | 17
  >=65 years | 0 | 3 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (17.35) | 50.8 (15.20) | 52.8 (13.40) | 51.3 (19.30) | 49.6 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 7
  Male | 1 | 9 | 3 | 2 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 10 | 4 | 3 | 20
  Asian | 0 | 1 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: AE tables are below in the Adverse Events section of this report.
Time Frame: week 52
Population: The Safety Analysis Set was comprised of all subjects that received study drug and with no protocol deviations having relevant impact on safety.
Measure: Count of Participants; unit: Participants
Groups:
- CGF166 Dose 30 μLEdit Single Dose Volume #2: single dose #2
- Total: Number of participants
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μLEdit Single Dose Volume #2 | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Participants | 3 | 6 | 4 | 3 | 16

2. Primary Outcome: Number of Adverse Events
Description: AE tables are below in the Adverse Events section of this report.
Time Frame: week 52
Population: as for outcome 1
Measure: Number; unit: Adverse events
Groups:
- Total: Number of AEs
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Adverse events | 9 | 16 | 13 | 8 | 46

3. Primary Outcome: Summary of Pure Tone Audiometry in Treated Ear Compared to Pretreatment Values
Description: Summary of pure tone audiometry air conduction thresholds at frequency 0.125 KHz
Time Frame: Days 29, 57, 85, 113, 141, 169, 358, 537, 600
Population: Pharmacodynamics (PD) analysis set was comprised of all subjects with any available PD data, who received any study drug and experienced no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: DECIBELS
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
DECIBELS
  Baseline | 63.3 (18.93) | 70.0 (14.62) | 70.0 (20.41) | 71.7 (16.07) | 69.3 (15.38)
  Day 29 | 61.7 (20.82) | 70.4 (22.10) | 85.0 (10.80) | 75.0 (15.00) | 72.5 (19.62)
  Day 57: number analyzed (Participants) | 3 | 11 | 4 | 3 | 21
  Day 57 | 61.7 (20.82) | 71.4 (15.34) | 86.3 (8.54) | 73.3 (15.28) | 73.1 (15.85)
  Day 85: number analyzed (Participants) | 3 | 4 | 4 | 3 | 14
  Day 85 | 61.7 (25.66) | 66.3 (14.36) | 88.8 (24.96) | 75.0 (15.00) | 73.6 (21.16)
  Day 113: number analyzed (Participants) | 3 | 11 | 4 | 3 | 21
  Day 113 | 60.0 (27.84) | 73.6 (14.33) | 92.5 (23.63) | 75.0 (15.00) | 75.5 (19.55)
  Day 141: number analyzed (Participants) | 3 | 4 | 4 | 3 | 14
  Day 141 | 60.0 (27.84) | 68.8 (14.93) | 91.3 (22.87) | 73.3 (14.43) | 74.3 (21.65)
  Day 169: number analyzed (Participants) | 0 | 7 | 0 | 2 | 9
  Day 169 |  | 72.1 (11.85) |  | 70.0 (7.07) | 71.7 (10.61)
  Day 358: number analyzed (Participants) | 0 | 4 | 0 | 2 | 6
  Day 358 |  | 80.0 (14.14) |  | 72.5 (10.61) | 77.5 (12.55)
  Day 537: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Day 537 |  | 82.5 (10.61) |  | 75.0 | 80.0 (8.66)
  Day 600: number analyzed (Participants) | 3 | 10 | 4 | 2 | 19
  Day 600 | 60.0 (27.84) | 77.5 (15.68) | 93.8 (9.46) | 82.5 (17.68) | 78.7 (18.77)

4. Primary Outcome: Summary Pure Tone Audiometry Bone Conduction Thresholds in Treated Ear by Time and Frequency
Description: Summary of pure tone audiometry bone conduction thresholds by time and frequency 0.250 KHz
Time Frame: Days 29, 57, 85, 113, 141, 169, 358,537, EoS
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
decibels
  Baseline | 55.0 (0.00) | 64.2 (28.83) | 87.5 (43.5) | 55.0 (0.00) | 65.9 (28.81)
  Day 29 | 55.0 (0.00) | 73.8 (31.49) | 63.8 (42.11) | 55.0 (0.00) | 66.8 (29.01)
  Day 57: number analyzed (Participants) | 3 | 11 | 4 | 3 | 21
  Day 57 | 50.0 (8.66) | 56.8 (7.83) | 90.0 (40.41) | 55.0 (0.00) | 61.9 (21.99)
  Day 85: number analyzed (Participants) | 3 | 4 | 4 | 3 | 14
  Day 85 | 48.3 (11.55) | 90.0 (40.41) | 90.0 (40.41) | 51.7 (5.77) | 72.9 (34.68)
  Day 113: number analyzed (Participants) | 3 | 11 | 4 | 3 | 21
  Day 113 | 50.0 (8.66) | 57.7 (23.17) | 86.3 (45.16) | 53.3 (2.89) | 61.4 (27.26)
  Day 141: number analyzed (Participants) | 3 | 4 | 4 | 3 | 14
  Day 141 | 46.7 (14.43) | 51.3 (7.50) | 90.0 (40.41) | 51.7 (5.77) | 61.4 (27.97)
  Day 169: number analyzed (Participants) | 3 | 7 | 0 | 2 | 9
  Day 169 | 0 (0) | 48.6 (8.52) |  | 50.0 (7.07) | 48.9 (7.82)
  Day 358: number analyzed (Participants) | 0 | 4 | 0 | 2 | 6
  Day 358 |  | 45.0 (8.16) |  | 55.00 (0.00) | 48.3 (8.16)
  Day 537: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3
  Day 537 |  | 50 (7.07) |  | 40 | 46.7 (7.64)
  End of Study: number analyzed (Participants) | 3 | 10 | 4 | 2 | 19
  End of Study | 48.3 (11.55) | 61.5 (22.37) | 90.0 (40.41) | 50.0 (7.07) | 64.2 (27.50)

5. Primary Outcome: Summary of Change From Baseline in Treated Ear's Pure Tone Audiometry Air Conduction Threshold by Frequency for Last Study Visit
Description: Summary of change from baseline in pure tone audiometry air conduction threshold by frequency for last study visit is presented in table below.
Time Frame: Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
decibels
  125 hz | -4.2 (9.46) | 6.7 (10.19) | 26.3 (17.02) | 5.0 (4.33) | 8.5 (13.88)
  250 Hz | -3.3 (6.29) | 6.0 (9.20) | 26.3 (26.65) | 0.8 (1.44) | 7.7 (15.52)
  500 Hz | 0 (5.00) | 7.7 (11.00) | 26.3 (23.32) | 0.8 (1.44) | 9.1 (14.91)
  1,000 Hz | -0.8 (3.82) | 8.1 (10.51) | 16.9 (8.98) | 5.8 (1.44) | 8.2 (9.89)
  2,000 Hz | 0.8 (6.29) | 6.0 (11.40) | 6.9 (8.51) | 0.8 (3.82) | 4.8 (9.48)
  3,000 Hz | 2.5 (2.50) | 5.8 (11.60) | 11.9 (11.06) | -4.2 (3.82) | 5.1 (10.59)
  4,000 Hz | 0.8 (1.44) | 4.4 (12.97) | 5.0 (4.08) | -0.8 (3.82) | 3.3 (9.83)
  6,000 Hz | 1.7 (2.89) | 3.3 (13.16) | 7.5 (15.00) | 1.7 (6.29) | 3.2 (11.60)
  8,000 Hz | 1.7 (2.89) | 2.9 (15.33) | -8.8 (17.50) | 4.2 (7.22) | 0.8 (13.94)

6. Primary Outcome: Summary of Change From Baseline in Non-treated Ear's Pure Tone Audiometry Air Conduction Threshold by Frequency for Last Study Visit
Description: Summary of change from baseline in Non-treated ear's pure tone audiometry air conduction threshold by frequency for last study visit is presented in table below.
Time Frame: Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
decibels
  125 hz | -2.5 (6.61) | 1.7 (4.92) | -3.1 (2.39) | -1.7 (3.82) | 8.5 (4.87)
  250 Hz | 0 (8.66) | 2.3 (5.48) | -2.5 (3.54) | 0.8 (2.89) | 7.7 (5.45)
  500 Hz | 0.8 (1.44) | 6.0 (18.87) | -2.5 (3.54) | -1.7 (2.50) | 9.1 (14.32)
  1,000 Hz | 1.7 (2.89) | 1.7 (4.81) | 0 (2.04) | -1.7 (1.44) | 8.2 (3.83)
  2,000 Hz | 0.8 (2.89) | 0.2 (7.27) | -0.6 (2.39) | -2.5 (4.33) | 4.8 (5.66)
  3,000 Hz | 0 (5.00) | 0.2 (4.94) | 0.6 (1.25) | -7.5 (2.50) | 5.1 (4.84)
  4,000 Hz | -2.5 (6.61) | 1.0 (3.76) | 1.3 (2.50) | -0.8 (6.29) | 3.3 (4.25)
  6,000 Hz | -0.8 (1.44) | -0.6 (3.56) | -8.1 (11.79) | -1.7 (5.77) | 3.2 (6.19)
  8,000 Hz | -3.3 (5.77) | -4.2 (10.78) | -8.8 (17.50) | -0.8 (6.29) | 0.8 (10.83)

7. Secondary Outcome: Number of Participants With Change in Brainstem Auditory Evoked Responses (BAER) Compared to Pretreatment Values
Description: BAERs was assessed with standard techniques for clinically significant threshold improvements compared to baseline levels.
Time Frame: 24 months
Population: PD analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Response in Vestibular Function in Treated Ear Compared to Pretreatment Values
Description: Response in vestibular assessments (Head impulse test (HIT), Vestibular evoked myogenic potential (VEMP), Subjective visual vertical (SVV)) to CGF166.
Time Frame: 24 months
Population: PD Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Changes in Auditory Functions (Speech Recognition) and Vestibular Functions Before and After IL Infusion of CGF166 Between the Study Ear and the Contralateral Ear
Description: Clinically signficant speech recognition improvement (word and/or sentence) following treatment. The individual auditory assessments were speech audiometry, AzBio sentence test, consonant nucleus consonant test, word recognition, Hearing-in-Noise Test (HINT), Brainstem auditory evoked response evaluations (BAER), Distortion product otoacoustic emission testing (DPOE) and shoebox audiometry.
Time Frame: 24 months
Population: PD analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total Number of participants
Arm/Group | CGF166 Dose 20 μL | CGF166 Dose 30 μL | CGF166 Dose 40 μL | CGF166 Dose 60 μL | Total
Number analyzed (Participants) | 3 | 12 | 4 | 3 | 22
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment until end of study treatment at 52 weeks
Description: AEs are any untoward sign or symptom that occurs during the study treatment
Groups:
- CGF166 20 μL: CCGF166X2201 20 μL
- CGF166 30 μL: CCGF166X2201 30 μL
- CGF166 40 μL: CCGF166X2201 40 μL
- CGF166 60 μL: CCGF166X2201 60 μL
Arm/Group | CGF166 20 μL | CGF166 30 μL | CGF166 40 μL | CGF166 60 μL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/12 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/12 | 4/4 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CGF166 20 μL (N=3) | CGF166 30 μL (N=12) | CGF166 40 μL (N=4) | CGF166 60 μL (N=3)
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 2 | 4 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Vestibular migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02132130/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02132130/SAP_001.pdf